CLINICAL TRIAL: NCT04607590
Title: Yoga Program for Couples Coping With Cancer
Brief Title: Yoga Program for Improving the Quality of Life in Couples Coping With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0887; NCI-2020-02943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0887 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-05-20; First posted 2020-10-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Carcinoma; Lung Carcinoma; Malignant Head and Neck Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Head and Neck Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (DY) (Experimental): Patients and their partners attend yoga sessions 3 days per week for up to 15 sessions, lasting 60 minutes each, in-person or via videoconferencing over the course of radiation therapy.
  Interventions: Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Yoga
- Group II (PY) (Experimental): Patients attend yoga sessions 3 days per week for up to 15 sessions, lasting 60 minutes each, in-person or via videoconferencing over the course of radiation therapy. Once data collection is completed, partners will be offered intervention materials, and encouraged to attend yoga classes at the Integrative Medicine Clinic.
  Interventions: Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Yoga
- Group III (WLC) (Experimental): Patients and their partners receive usual care. Once data collection is completed, couples may participate in the DY or PY program of their choice over 60 minutes each. Partners are also offered intervention materials along with five 60 minute optional yoga sessions.
  Interventions: Other: Best Practice; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Yoga

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group III (WLC)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Yoga — Participate in yoga sessions
  Other Names: Yoga Therapy

SUMMARY:
This clinical trial seeks to learn if a yoga program can improve physical performance, quality of life and symptom burden in cancer patients who are undergoing radiation therapy, and their partners. Taking part in yoga or stretching sessions may lower distress, improve quality of life, and/or may improve sleep and fatigue for cancer patients and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the extent to which the dyadic yoga (DY) program improves patient objective physical performance as compared to the waitlist control (WLC) group (primary comparison) and the patient-only yoga (PY) group (exploratory comparison).

SECONDARY OBJECTIVE:

I. To examine the extent to which the DY program improves patient and partner quality of life (QOL) compared to the WLC group (primary comparison) and the PY group (exploratory comparison).

TERTIARY OBJECTIVE:

I. To examine the extent to which the DY program reduces patient healthcare utilization (i.e., emergency room visits, hospital admissions, and feeding tube insertions) and patient and partner work productivity compared to the WLC group (primary comparison) and the PY group (exploratory comparison).

EXPLORATORY OBJECTIVE:

I. To explore if, compared to the WLC and PY groups, the DY program improves symptom burden and symptom management skills at the end of treatment, which will in turn mediate intervention outcomes at the subsequent follow-up assessments.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I (DY): Patients and their partners attend yoga sessions 3 days per week for up to 15 sessions, lasting 60 minutes each, in-person or via videoconferencing over the course of radiation therapy.

GROUP II (PY): Patients attend yoga sessions 3 days per week for up to 15 sessions, lasting 60 minutes each, in-person or via videoconferencing over the course of radiation therapy. Once data collection is completed, partners are offered intervention materials, and encouraged to attend yoga classes at the Integrative Medicine Clinic.

GROUP III (WLC): Patients and their partner receive usual care. Once data collection is completed, couples may participate in the DY or PY program of their choice over 60 minutes each. Partners are also offered intervention materials along with five 60 minute optional yoga sessions.

After completion of radiation therapy, patients are followed up at 1 , 2, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS ONLY: Diagnosed with a lung cancer, head and neck cancer, or esophageal cancer to receive at least 25 fractions over 5 weeks of radiation therapy (RT)
* PATIENTS ONLY: Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* PATIENTS ONLY: Having a spouse or cohabitating partner (same or opposite sex) willing to participate
* PATIENTS AND PARTNERS: Must be at least 18 years old
* PATIENTS AND PARTNERS: Must be able to read and speak English
* PATIENTS AND PARTNERS: Must be able to provide informed consent

Exclusion Criteria:

* PATIENTS ONLY: Who have regularly (self-defined) participated in a mind-body practice or exercise program in the year prior to diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
The patient 6-minute walk test (6-MWT) over the 6-month follow up (6-MFU) | At the 3-month follow-up
  This analysis will be imbedded in a linear mixed-effects (alternatively known as the multilevel) modeling (MLM) analysis, with repeated measures over time (i.e., at end of treatment, 3- and 6-month follow-ups). Potential interaction terms will be included and tested, in particular, between the intervention and time. The repeated measures correlation structure will be selected using the Bayesian information criterion (BIC). The difference between dyadic yoga (DY) and waitlist control (WLC) at 3MFU is considered the primary and confirmatory comparison and will be tested at a two-sided 0.025 significance level. Additionally, on an exploratory basis, will conduct an omnibus test on the overall differences in 6MWT across the three groups at 3-month follow-up, as well as pairwise comparisons between the patient yoga (PY) and WLC and between DY and PY. Exploratory comparisons will be primarily interpreted based on clinically significant difference, which is 70m for the study population.

SECONDARY OUTCOMES:
Patient and partner short form survey (SF-36) domains | At each follow-up time point (1 month follow-up to 6-month follow-up)
  Analyses will be similar to those for the primary outcome, except that will use a dyadic model assuming additional dependence in outcomes between patient and partner outcomes. Repeated measures over time will include at the end of treatment, 1-, 3- and 6-month follow-ups. Will examine the individual SF-36 domains as well as the physical (PCS) and mental component summaries (MCS). Patient and partner overall quality of life (QOL) will be measured with the Medical Outcomes Study 36-item short-form survey (SF-36) assessing 8 distinct domains: physical functioning, physical impediments to role functioning, pain, general health perceptions, vitality, social functioning, emotional impediments to role functioning, and mental health. The SF-36 will take up to 7 minutes to complete and will be assessed at each follow-up time point (time point 1 [T1] - time point 6 [T6]).

OTHER OUTCOMES:
Healthcare utilization and work productivity | During radiation therapy (RT) and 90-days post-RT (T1-T5)
  To assess the differences between groups in patient healthcare utilization will test the patient emergency department (ED) visits, hospital admissions (HA) admissions and feeding tube (FT) insertions. Will use a Chi-squared or Fisher's exact test, as appropriate, to compare the probability of healthcare services using a binary outcome (yes/no) between groups at a two-sided 0.025 significance level. Additional analyses will examine the number of times a patient visited the ED during the specified period. As a follow-up analysis, will examine group differences with logistic regression using randomization factors as model covariates (i.e., age, sex, ethnicity, stage, smoking status) as these factors may be associated with the study outcomes. Productivity loss will be measured by the Work Productivity and Activity Impairment General Health (WPAI-GH) assessing presence at the work place. Both patients and partners will complete items pertaining to productivity loss due to their health.
Physical and emotional intimacy | Baseline, end of treatment (T3), 3 months after RT (T5) and 6 months after RT (T6)
  Sexual problems will be assessed with Majerovitz and Revenson's 6-item measure of sexual problems, which have successfully been used in our previous research in couples coping with cancer. Emotional intimacy will be measures with the validated and frequently used 6-item Personal Assessment of Intimacy in Relationships (PAIR) instrument, which has been validated in cancer. Will explore if the DY intervention improves physical and emotional intimacy following the procedures as described for the QOL (secondary) outcome. Will control for values of outcomes at baseline, as well as the randomization factors, in all the above analyses to improve power of the comparisons.
Treatment efficacy | At the end of radiation therapy (T2)
  Will examine if treatment efficacy on outcomes measured at 3MFU (T4) are achieved through improved symptoms and symptom management skills at the end of RT (T2) using linear regression analysis in both the intervention-mediator: (a) and intervention plus (+) mediator-outcome (b) paths. Ninety-five percent Bootstrap confidence intervals (CIs) will be constructed to assess the significance of the indirect (or mediation) effects defined using the product-of-coefficient approach. Will also use multilevel modeling (MLM) to test for interaction effects between intervention and the priori moderators, baseline depressive symptoms and dyadic adjustment. Significant interactions will be probed using simple slope analyses following the procedure developed for multilevel modeling by Preacher, Curran, and Bauer. These analyses will use a two-sided 0.05 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org